CLINICAL TRIAL: NCT07215650
Title: A Phase 1b, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Patients With Generalized Myasthenia Gravis (gMG)
Brief Title: Clinical Study of Cizutamig in Generalized Myasthenia Gravis (gMG)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Candid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND106-107
Record Dates: First submitted 2025-09-24; First posted 2025-10-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cizutamig (Experimental)
  Interventions: Drug: Cizutamig

INTERVENTIONS:
Drug: Cizutamig — Cizutamig will be dosed according to the protocol
  Other Names: CND106

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK, PD, immunogenicity, and preliminary clinical activity of Cizutamig in patients with Generalized Myasthenia Gravis.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary clinical activity of cizutamig in patients with Generalized Myasthenia Gravis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old at the time of signing the Informed Consent Form (ICF);
2. Diagnosed with MG, classified as MGFA Class II-IVa, and judged by the investigator as unlikely to require respiratory support during the study;
3. At screening, the Myasthenia Gravis Activities of Daily Living (MG-ADL) score ≥ 5, with non-ocular items accounting for ≥ 50% of the total score, and GMG ≥ 11;
4. Inadequate response to conventional therapies or lack of effective treatment options, defined as disease recurrence or progression despite treatment with corticosteroids, immunosuppressants (e.g., azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine A, methotrexate), or biologics (e.g., rituximab), and/or lack of effective treatment methods.

Exclusion Criteria:

1. Any history of CAR-T or TCE therapy targeting any antigen or BCMA-targeted therapy;
2. Use of any approved immunosuppressive drugs not listed here within 12 weeks or 5 half-lives (whichever is longer) before screening, unless approved by the medical monitor;
3. Participation in any investigational trial involving non-biological agents within 4 weeks or 5 half-lives (whichever is longer) of the investigational product (IP) before screening;
4. Participation in any investigational trial involving biological agents within 12 weeks or 5 half-lives (whichever is longer) of the IP before screening;
5. Administration of live vaccines within 4 weeks before screening;
6. History of progressive multifocal leukoencephalopathy;
7. History of primary immunodeficiency (e.g., hypogammaglobulinemia) or hereditary complement deficiency;
8. Presence of one or more significant concurrent diseases, as judged by the investigator, including but not limited to:

   1. Poorly controlled diabetes
   2. Chronic kidney disease stages IIIb, IV, or V
   3. Severe chronic pulmonary disease (e.g., requiring supplemental oxygen) or respiratory failure
9. Any severe medical condition or clinically significant laboratory abnormality that, in the judgment of the investigator or medical monitor, would compromise the patient's safe participation and completion of the study or may affect protocol compliance or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events through end of study | Baseline to Month 12
Changes from baseline in vital signs through end of study: body temperature | Baseline to Month 12
Changes from baseline in vital signs through end of study: heart rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: respiratory rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: blood pressure | Baseline to Month 12
Changes from baseline in vital signs through end of study: pulse oximetry | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: PR interval | Baseline to Month12
Changes from baseline in ECG parameters through end of study: QRS interval | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: QTcF interval | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: serum chemistry | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: hematology | Baseline to Month 12

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters for Cizutamig: Cmax | Baseline to Month 12
PK parameters for Cizutamig: time of maximum concentration | Baseline to Month 12
PK parameters for Cizutamig: area under the concentration-time curve | Baseline to Month 12
PK parameters for Cizutamig: clearance | Baseline to Month 12
PK parameters for Cizutamig: volume of distribution | Baseline to Month 12
PK parameters for Cizutamig: half-life | Baseline to Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No